CLINICAL TRIAL: NCT05768256
Title: A Study of Treatment Efficacy of Mindfulness-based Cognitive Therapy for Distress (MBCT-D) in Advanced Cancer Patients Using Neurophysiological Data
Brief Title: Treatment Efficacy of Mindfulness-based Cognitive Therapy for Distress in Advanced Cancer Patients
Acronym: MBCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: CHA University (Other)
Responsible Party: Principal Investigator, Chun Il Park, Associate Professor, CHA University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHAMC 2022-12-050; NRF-2021R1I1A1A01048880 (Other Grant/Funding Number: Ministry of Education)
Record Dates: First submitted 2023-02-07; First posted 2023-03-14 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Cancer Pain; Cancer; Distress, Emotional; Therapy-Associated Cancer; Psychiatric or Mood Diseases or Conditions; Psychological Distress
MeSH Terms: conditions — Cancer Pain; Neoplasms; Neoplasms, Second Primary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Advanced cancer patients (Experimental)
  Interventions: Behavioral: Mindfulness-Based Cognitive-behavioral Therapy for Distress

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive-behavioral Therapy for Distress — Mindfulness-based cognitive-behavioral therapy, MBCT, is a modified form of cognitive-behavioral therapy that incorporates mindfulness practices that include present moment awareness, meditation, and breathing exercises. Advanced cancer patients will participate in the study until the end of the study (Feb 2024). After registering for the study, the study subjects receive mindfulness-based cognitive behavioral therapy once a week for eight weeks.

SUMMARY:
'Distress' refers to emotional distress, including psychological distress, in cancer patients. This study aims to explore whether mindfulness-based cognitive-behavioral therapy for cancer patients is effective in relieving distress and to discover neurophysiological factors that contribute to relieving distress. Mindfulness meditation, which is the core of mindfulness-based cognitive behavioral therapy, can develop cognitive flexibility through 'awareness of what is happening now'. In this study, a mindfulness-based cognitive behavioral therapy program is implemented for patients with advanced cancer, and clinical characteristics and conditions including distress level are observed through questionnaires and interviews. In addition, genetic data and brain imaging data are collected through blood sampling and brain magnetic resonance imaging. The ultimate goal of this study is to prove the therapeutic efficacy of a mindfulness-based cognitive behavioral therapy program for distress of patients with advanced cancer through an in-depth and multifaceted integrated approach, and to understand the related neurophysiological mechanisms.

DETAILED DESCRIPTION:
The number of subjects participating in this study is up to 40 advanced cancer patients. The research subject is responsible for the medical expenses incurred in the usual standard medical procedures, and the researcher is responsible for the examination expenses (brain magnetic resonance imaging, blood sampling) performed by participating in other studies.

This study runs until Feb 01, 2024. After enrolling in the study, patients with advanced cancer participate in mindfulness-based behavioral therapy once a week for eight weeks. All research subjects participating in this study will have an interview to collect basic information, fill out a questionnaire for index evaluation, blood collection, and brain magnetic resonance imaging. Participants participating in this study will receive specific evaluations as follows.

1. Interview to gather basic information: demographic information, (if applicable) psychiatric symptoms and treatment-related information are collected.
2. Filling out questionnaires for psychological evaluation and behavioral data collection: 4 times [Baseline, 2 weeks later, 4 weeks later, 8 weeks later (Post-treatment)], Psychiatry Fill out a questionnaire to comprehensively evaluate your symptoms and psychological state.
3. Blood collection: 6ml of blood is collected twice before and after treatment.
4. Brain Magnetic Resonance Imaging: Make an appointment and visit the examination room in the hospital to perform a total of 2 times before and after treatment.

Clinical symptom and progress data are collected if patients have previously been treated at this hospital, and medical information that occurs after study registration is collected every one month during the study participation period.

Distress Indicators

* 2022 NCCN Guidelines for Distress Management's Korean version of Distress Thermometer (DT) and Problem List (PL)
* Perceived Stress Scale-4 (PSS-4) Indicators of depression and anxiety characteristics
* Brief Edinburgh Depression Scale (BEDS)
* Beck Depression Inventory-ll (BDI-ll)
* Beck Anxiety Inventory (BAI)
* Hospital Anxiety and Depression Scale (HADS) Mindfulness Characteristics and Symptom Related Indicators
* Toronto Mindfulness Scale (TMS)
* Self-Compassion Scale-Short Form (SCS-SF)
* Demoralization Scale-II (DS-II-Kr)
* Thought-Action Fusion Scale (TAFS) Quality of life and resilience indicators
* Functional Assessment Cancer Therapy-General (FACT-G)
* WHO Quality of Life-BREF (WHOQOL-BREF)
* The Brief Resilience Scale (BRS) Epigenetic data
* DNA methylation analysis flow DNA preparation → uracil change of non-methylated cytosine using bisulfate → amplification using PCR → methylation detection by methylation specific PCR
* Selection of candidate genes - Experience in prior research on OXTR and FKBP5gene → Application to same gene methylation studies Brain imaging data
* Acquisition of magnetic resonance imaging (MRI) - structural imaging (T1), functional imaging (fMRI), diffusion tensor imaging (DTI)

ELIGIBILITY:
Inclusion Criteria:

* A person diagnosed with gastric cancer, colon cancer, lung cancer, liver cancer, breast cancer, cervical cancer, prostate cancer, or other cancers from a doctor, and a advanced cancer patient with a cancer stage of 2 to 4
* Those who wish to participate in the Mindfulness-Based Cognitive Behavioral Treatment for distress (MBCT-D) program

Exclusion Criteria:

* A person with a history of neurological disease, head trauma accompanied by loss of consciousness, brain metastasis of cancer, and mental retardation (IQ<70).
* Pregnant and lactating
* If the symptoms are severe or the reality testing ability and judgment are considered to be significantly deteriorated through a mental health examination by a psychiatrist
* A person who is determined to be at risk of serious suicide or violent behavior in the mental state test
* A foreigner (a non-Korean person)
* A person who is illiterate in Korean
* A left-handed person
* A person who has previously experienced mindfulness-based cognitive behavioral therapy
* A person who the researcher determines that it is inappropriate to participate in clinical research for other reasons

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Distress level change | at baseline, 2nd week, 4th week, 8th week
  Measure the distress levels using the Distress Thermometer. The Distress Thermometer ranged from 0 to 10. Higher scores indicate more severe distress.
Gray matter volume change | at baseline, 8th week
  Measure the gray matter volume using fast spoiled gradient-echo (FSPGR) of three-dimensional brain Magnetic Resonance Imaging data.
Gray matter thickness change | at baseline, 8th week
  Measure the gray matter thickness using fast spoiled gradient-echo (FSPGR) of three-dimensional brain Magnetic Resonance Imaging data.
White matter microstructure change | at baseline, 8th week
  Measure the white matter microstructure using diffusion tensor imaging (DTI) of three-dimensional brain Magnetic Resonance Imaging data.
Brain functional connectivity change | at baseline, 8th week
  Measure the functional connectivity using functional magnetic resonance imaging (fMRI) of three-dimensional brain Magnetic Resonance Imaging data.
DNA methylation levels change | at baseline, 8th week
  Measure the DNA methylation levels using blood collection.

SECONDARY OUTCOMES:
Depression level change | at baseline, 2nd week, 4th week, 8th week
  Measure the depressive levels using the Brief Edinburgh Depression Scale. The Brief Edinburgh Depression Scale ranged from 0 to 18, with higher scores indicating more depression.
Depression level change | at baseline, 2nd week, 4th week, 8th week
  Measure the depressive levels using the Beck Depression Inventory-ll. The Beck Depression Inventory-ll ranged from 0 to 63, with higher scores indicating more depression.
Depression level change | at baseline, 2nd week, 4th week, 8th week
  Measure the depressive levels using the Hospital Anxiety and Depression Scale. The Hospital Anxiety and Depression Scale ranged from 0 to 21, with higher scores indicating more depression.
Anxiety level change | at baseline, 2nd week, 4th week, 8th week
  Measure the depressive levels using the Hospital Anxiety and Depression Scale. The Hospital Anxiety and Depression Scale ranged from 0 to 21, with higher scores indicating more anxiety.
Anxiety level change | at baseline, 2nd week, 4th week, 8th week
  Measure the anxiety levels using the Beck Anxiety Inventory. Scale ranged from 0 to 63, with higher scores indicating more anxiety.
Mindfulness level change | at baseline, 2nd week, 4th week, 8th week
  Measure the mindfulness levels using the Toronto Mindfulness Scale. The Toronto Mindfulness Scale ranged from 13 to 65, with higher scores indicating more mindfulness.
Self-compassion level change | at baseline, 2nd week, 4th week, 8th week
  Measure the mindfulness levels using the Self-Compassion Scale-Short Form. The Self-Compassion Scale-Short Form ranged from 12 to 60, with higher scores indicating more self-compassion.
Demoralization level change | at baseline, 2nd week, 4th week, 8th week
  Measure the mindfulness levels using the Demoralization Scale-II. The Demoralization Scale-II ranged from 0 to 32, with higher scores indicating more demoralization.
Thought-action fusion level change | at baseline, 2nd week, 4th week, 8th week
  Measure the mindfulness levels using the Thought-Action Fusion Scale. The Thought-Action Fusion Scale ranged from 0 to 76, with higher scores indicating a greater thought-action fusion.
Health-related quality of life level change | at baseline, 2nd week, 4th week, 8th week
  Measure the health-related quality of life levels using the Functional Assessment Cancer Therapy-General. The Functional Assessment Cancer Therapy-General ranged from 0 to 108, with higher scores indicating more health-related quality of life.
Physical-related quality of life level change | at baseline, 2nd week, 4th week, 8th week
  Measure the physical-related quality of life levels using the Physical domain of WHO Quality of Life-BREF. The Physical domain of WHO Quality of Life-BREF ranged from 0 to 20, with higher scores indicating more physical-related quality of life.
Psychological-related quality of life level change | at baseline, 2nd week, 4th week, 8th week
  Measure the psychological-related quality of life levels using the Psychological domain of WHO Quality of Life-BREF. The Psychological domain of WHO Quality of life-BREF ranged from 0 to 20, with higher scores indicating more psychological-related quality of life.
Social-related quality of life level change | at baseline, 2nd week, 4th week, 8th week
  Measure the social-related quality of life levels using the Social domain of WHO Quality of Life-BREF. The Social domain of WHO Quality of life-BREF ranged from 0 to 20, with higher scores indicating more social-related quality of life.
Environmental-related quality of life level change | at baseline, 2nd week, 4th week, 8th week
  Measure the environmental-related quality of life levels using the Environmental domain of WHO Quality of Life-BREF. The Environmental domain of WHO Quality of Life-BREF ranged from 0 to 20, with higher scores indicating more environmental-related quality of life.
Resilience level change | at baseline, 2nd week, 4th week, 8th week
  Measure the resilience levels using the The Brief Resilience Scale. The Brief Resilience Scale ranged from 6 to 30, with higher scores indicating more resilience.

CONTACTS AND LOCATIONS:
Locations (1):
- CHA Bundang Medical Center, Seongnam-si, Kyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wurtzen H, Dalton SO, Elsass P, Sumbundu AD, Steding-Jensen M, Karlsen RV, Andersen KK, Flyger HL, Pedersen AE, Johansen C. Mindfulness significantly reduces self-reported levels of anxiety and depression: results of a randomised controlled trial among 336 Danish women treated for stage I-III breast cancer. Eur J Cancer. 2013 Apr;49(6):1365-73. doi: 10.1016/j.ejca.2012.10.030. Epub 2012 Dec 19. PMID 23265707
- [Background] Kim B, Lee SH, Kim YW, Choi TK, Yook K, Suh SY, Cho SJ, Yook KH. Effectiveness of a mindfulness-based cognitive therapy program as an adjunct to pharmacotherapy in patients with panic disorder. J Anxiety Disord. 2010 Aug;24(6):590-5. doi: 10.1016/j.janxdis.2010.03.019. Epub 2010 Apr 3. PMID 20427148